CLINICAL TRIAL: NCT05136105
Title: Preventing Trauma Symptoms in the Aftermath of Sexual Abuse in Children and Adolescents in Burundi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal Investigator, University of Konstanz
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UKAC2021
Record Dates: First submitted 2021-11-12; First posted 2021-11-26 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Posttraumatic Stress Disorder; Mental Health Issue; Family Dynamics
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Two cohorts. The first cohort receiving treatment as usual in Burundi, mostly a waiting control group, the second cohort receiving a three session family focused intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventive Narrative Exposure Therapy (PreNET) family intervention (Experimental): The intervention group receives treatment as usual in the first aid center for survivors of sexual abuse. This includes medical and judicial assistance if necessary. Furthermore, they receive the psychological family focused intervention.
  The intervention consists of a total of three sessions with the aim of reestablishing and validating the relationship between sexually abused children and their parents. The intervention focuses on psychoeducation regarding shame and other trauma related disorders. Further, the acknowledgement of shame and embarrassment as well as parental skills are intended to be improved.
  Interventions: Behavioral: Preventive Narrative Exposure Therapy (PreNET) family intervention
- No Intervention group (No Intervention): The control group will receive only the assessments, and treatment as usual in a first aid center for survivors of sexual abuse. This includes usually a brief assessment of what happened as well as medical and judicial assistance if necessary.

INTERVENTIONS:
Behavioral: Preventive Narrative Exposure Therapy (PreNET) family intervention — Sessions: (1) Participants are invited to narrate the event in detail, in line with the protocol of the trauma-focused intervention NET. Furthermore, participants and caregiver(s) will receive a brief psychoeducation about expected symptoms and supportive behaviour in the aftermath of sexual violence.
  (2) Two weeks after session 1, the second session focuses on caregiver only and their emotions. The narration of the event is read to the caregiver(s). Caregiver(s) receive assistance regulating their emotions. They receive psychoeducation on how to support their child.
  (3) Two weeks after the second session, the children assisted by their caregivers lay a chronological lifeline of their most important life experiences. The chronology and the context of the traumatic events is reinforced. The narration of the sexual abuse is read again to the child and the caregiver(s). The caregiver(s) are encouraged to support emotionally their child during the renarration.
  Arms: Preventive Narrative Exposure Therapy (PreNET) family intervention

SUMMARY:
Survivors of sexual violence are particularly vulnerable to develop psychological as well as physical health problems, Burundian children and adolescents being at elevated risk. Psychosocial care, and trauma-focused interventions, nevertheless, are near absent in Burundi.

The purpose of this project is to ameliorate psychosocial care for survivors of sexual violence in strengthening health care competencies by implementing evidence-based intervention strategies. We intend to develop an approach identifying particularly vulnerable children and adolescents and testing a preventive family-oriented psychotherapeutic approach. The latter aims at reducing stigmatization and at promoting the processing of the event within families. The project involves two cohorts, which are assessed enrolling them in the study, during a three-months and a 12-months follow-up.

DETAILED DESCRIPTION:
Survivors of sexual violence are particularly vulnerable to develop psychological as well as physical health problems, children and adolescents being at particular risk. Residing in conflict zones with disrupted community structures and social norms, substantially increases the risk for interpersonal violence, especially sexual abuse. The post-war country Burundi shows high prevalence rates for childhood sexual abuse. Adequate psychosocial care and trauma-focused interventions, however, are near absent, especially in rural areas.

Furthermore, talking about sexual activities remains a taboo-topic in Burundi, and particularly talking about sexual abuse. Survivors often suffer from stigmatization and therefore conceal their abusive experience. Recent studies, however, accentuate the importance of social support, notably parental acceptance, in the aftermath of sexual abuse. Parental acceptance shows buffering effects of sequelae following sexual abuse. Conversely, parental rejection, especially coming from the father, lowers the self-esteem and leads to emotional unresponsiveness and negative self-cognitions. Rejection thus risks to exacerbate feelings of shame and the internalization of stigma. Hence, the implementation of family-oriented interventions is crucial for effective treatment outcomes.

The purpose of this project is thus to ameliorate psychosocial care for survivors of sexual violence in strengthening health care competencies by implementing evidence-based intervention strategies. Combining insights from the aforementioned research, cognitive behavioural strategies, and cultural aspects we developed a preventive treatment approach aiming to address (1) the building block effect using trauma-therapeutic methods, (2) social exclusion by family members and society, and (3) communication about the incident and associated emotions within the family. The intervention consisted of three sessions. The first cohort included in the study does not receive the intervention in order to establish a baseline assessment of the course of mental health symptoms in the aftermath of sexual violence, and to help identify those in need of psychosocial assistance. The second cohort is offered the family intervention.

Follow-up assessments are planned at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Sexual abuse within the past month
* Participants are recruited when they approach a first aid center for survivors of sexual abuse

Exclusion Criteria:

* Psychotic symptoms
* Cognitive disability
* Current use of mind altering drugs

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
1. Change in mental health measured via the Strengths and Difficulties Questionnaire (SDQ) | baseline; 3-month follow-up; 12-months follow-up
  25 items, 5 subscales (conduct problems, hyperreactivity, emotional symptoms, peer problems, pro-social behavior), answer categories: 0 (not true) - 2 (certainly true). Subscale scores ranging from 0 - 10, overall score ranges from 0 - 40.
2. Change in PTSD symptom severity measured via the University of California in Los Angeles(UCLA)-PTSD Reaction Index | 3-month follow-up; 12-months follow-up
  27 items (DSM-5 diagnostic criteria for PTSD); answer categories frequency scored: 0 (none of the time) - 4 (all of the time). Overall score ranges from 0 - 80.

SECONDARY OUTCOMES:
3. Change in abuse-related parental acceptance-rejection | 3-month follow-up; 12-months follow-up
  Parental Acceptance and Rejection Questionnaire, short form; 24 items ranging from 1 - 4. Overall score ranges from 24 - 96.

CONTACTS AND LOCATIONS:
Locations (1):
- vivo international & Psychologues sans Frontières mental health center, Bujumbura, Bujumbura Mairie Province, Burundi

REFERENCES:
- [Derived] Schneider J, Rukundo-Zeller AC, Bambonye M, Muhoza JA, Ndayikengurukiye T, Nitanga L, Rushoza AA, Crombach A. Preventing Childhood Sexual Abuse Related Mental Health Deterioration Using a Narrative Family Intervention in Burundi. Res Child Adolesc Psychopathol. 2025 Jul;53(7):1061-1076. doi: 10.1007/s10802-025-01328-8. Epub 2025 May 10. PMID 40347425